CLINICAL TRIAL: NCT06755177
Title: Be Cautious of the Endogenous Endophthalmitis--Clinical Characteristics and Visual Prognosis of 104 Cases of Infectious Endophthalmitis
Brief Title: Clinical Features and Visual Prognosis of Infectious Endophthalmitis
Status: Completed | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024112001
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-10

CONDITIONS: Endophthalmitis
Keywords: Infectious endophthalmitis; Endogenous endophthalmitis; Exogenous endophthalmitis
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this observational study was to retrospectively examine the clinical data of patients with infectious endophthalmitis and to analyse their clinical characteristics.

The main question it aims to answer is: to find the differences between endogenous and exogenous endophthalmitis and to provide new ideas for the diagnosis and treatment of infectious endophthalmitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with infectious endophthalmitis by specialist examination. The clinical diagnosis of endophthalmitis was established on the basis of clinical signs and symptoms, including ocular pain, loss of vision, eyelid oedema, conjunctival congestion, inflammation of the anterior chamber (flare-ups, cells, pupillary fibrin membranes, and pus accumulation in the anterior chamber), vitritis, and vitreous clouding on B-scan ultrasound. The diagnosis of infectious endophthalmitis was clarified by the aqueous vitreous pathogen detection test.

Exclusion Criteria:

* Patients with incomplete medical records; non-infectious uveitis, retinal tumour disease, ocular ischaemia syndrome and other diseases with similar manifestations to endophthalmitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inhabitants
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-11 (Actual)

PRIMARY OUTCOMES:
visual acuity | Pre-operative, post-operative follow-up at 1 month, 3 months, 1 year, etc.
  best-corrected visual acuity （BCVA）

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No